CLINICAL TRIAL: NCT00000322
Title: Tyrosine for Methamphetamine Dependence
Brief Title: Tyrosine for Methamphetamine Dependence - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-10739-1; R01-10739-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1997-04

CONDITIONS: Amphetamine-Related Disorders
Keywords: amphetamine dependence
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — Tyrosine

INTERVENTIONS:
Behavioral: Tyrosine

SUMMARY:
The purpose of this study is to evaluate efficacy of tyrosine as a treatment for methamphetamine dependence in an outpatient treatment setting providing group psychosocial interventions. Examine effect of tyrosine on abstinence, retention in treatment, and craving."

DETAILED DESCRIPTION:
Evaluate efficacy of tyrosine as a treatment for methamphetamine dependence in an outpatient treatment setting providing group psychosocial interventions. Examine effect of tyrosine on abstinence, retention in treatment and craving.

ELIGIBILITY:
Inclusion Criteria:

18-65 years of age. Able to provide informed consent. Desire to reduce/eliminate methamphetamine use. Used within the past two weeks. Meet DSM criteria for methamphetamine dependence.

Exclusion Criteria:

No dependence (within the past 12 months) for other durgs except nicotine. No history or family history of tyrosine intolerance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89
Dates: Start 1997-04; Study Completion 2001-12

PRIMARY OUTCOMES:
Craving
Drug use
Retention
Functioning

CONTACTS AND LOCATIONS:
Overall Officials: Gantt Galloway, Pharm.D., Principal Investigator — Haight Ashbury Free Clinics
Locations (1):
- Haight Ashbury Free Clinics, San Francisco, California, United States